CLINICAL TRIAL: NCT01961648
Title: Effect of Increasing Respiratory Drive on Severity of Obstructive Apnea
Brief Title: Respiratory Drive on Obstructive Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators were not able to continue recruiting and enrolling.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2012:132
Record Dates: First submitted 2013-09-06; First posted 2013-10-11 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2013-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Apnea; Sleep Apnea Disorder; Respiratory chemical drive; CO2
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea | interventions — Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dead space (Active Comparator): Participant will sleep connected to a mask with added dead space half of the night
  Interventions: Device: Rebreathing bag; Device: Mask
- room air (Sham Comparator): Participant will sleep connected to a mask open to rrom air, half of the night
  Interventions: Device: Sham rebreathing; Device: Mask

INTERVENTIONS:
Device: Rebreathing bag
  Other Names: CO2 rebreathing; Dead space
  Arms: Dead space
Device: Sham rebreathing
  Other Names: Room air
  Arms: room air
Device: Mask

SUMMARY:
This study is being conducted to determine whether inhaling exhaled carbon dioxide is effective for the treatment of sleep apnea. A mild increase in this gas can stimulate the respiratory drive by 2-3 fold, which in turn can stimulate the upper airway dilator muscles and decrease the severity of obstructive sleep apnea by at least 50% in selected patients.

DETAILED DESCRIPTION:
During wakefulness pharyngeal dilator muscles (dilators) provide the necessary force to permit an adequate flow in all subjects regardless of how collapsible their passive pharynx is. This dilator activity is substantially lost at sleep onset. Subjects in whom the passive pharynx cannot permit adequate ventilation must recruit dilators through reflex mechanisms if they are to remain asleep. Dilators can be recruited reflexly via changes in blood gas tensions and in afferent activity of pharyngeal mechanoreceptors.

Patients with obstructive sleep apnea (OSA) develop repetitive obstructive events during which air flow decreases substantially (hypopneas) or ceases altogether (apneas). These last from 10 to >60 seconds following which there is a substantial increase in ventilation (hyperventilatory phase) that lasts for several breaths. The cycle then repeats. Arousal from sleep occurs at some point during the hyperventilatory phase in the vast majority of obstructive respiratory events. However it has been shown that in the majority of OSA patients, the reflex mechanisms are competent and can deal with the obstruction without arousal. The respiratory drive must increase a finite amount before the upper airway muscles begin responding to increasing respiratory drive, and often the patient wakes up first. Thus, when a subject with a narrowed or more compliant pharynx falls asleep and obstructs his/her airway, blood gas tensions must deteriorate a threshold amount before the pharyngeal dilators begin responding. Once this threshold is reached, the dilators respond briskly to further changes in blood gas tensions and open the airway. This threshold was termed the Effective Recruitment Threshold (TER).

The basis for this research project is that if respiratory drive can be maintained at or near the threshold, the dilators would respond promptly to any obstruction and there would be little further increase in respiratory drive during obstruction.We estimate that the required increase in drive can be attained by simply raising carbon dioxide pressure (PCO2) 2-3 mmHg, a highly tolerable increase. We intend to increase respiratory drive on a continuous basis, beginning before sleep by asking the participants to breath through a regular continuous positive airway pressure (CPAP) mask with added dead space.

To increase dead-space we will modify commercial rebreathing bags used for oxygen therapy so that the amount of rebreathing can be adjustable. This should raise arterial carbon dioxide pressure (PaCO2) a few millimetres of mercury (mmHg) in the steady state. Upon sleep, the respiratory drive would be at or above TER in nearly half the patients. Should the airway obstruct, the dilator muscles would be in a position to respond promptly, preventing an acute further rise in respiratory drive. This will reduce the frequency of obstructive respiratory events by >50% in at least half the patients, and improve sleep quality and nocturnal oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe OSA Apnea Hypopnea Index > 20/hr.
* Minimum oxygen saturation by pulse oximetry (SpO2) during events >70% throughout sleep during the clinical sleep study

Exclusion Criteria:

* Neuromuscular disease.
* Obesity-hypoventilation syndrome.
* Chronic obstructive pulmonary disease.
* Pregnancy.
* Significant comorbidities:

  1. Dialysis-dependant renal failure
  2. Severe asthma
  3. Congestive
  4. Heart failure
  5. Previous stroke
* Recent (within 3 months) myocardial infarction or Active coronary ischemia event.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total Apnea-hypopnea index (AHI) | Eight to ten hours. Within the same study night, the AHI will be compared at baseline and at the end of the intervention period
  We expect that at least half the patients will undergo >50% reduction in their AHI relative to the control part of the study. The baseline apnea-hypopnea index will be established during the sham intervention, and will be compared to the AHI at the end of the CO2 rebreathing intervention.

SECONDARY OUTCOMES:
Sleep quality as assessed by Total Sleep Time. Sleep Efficiency, and Arousal Index | Eight to ten hours. Within the same study night, the sleep quality conventional measurements will be compared at baseline and at the end of the intervention period
  The sleep architecture assessed by the sleep efficiency, number of arousals and awakenings, and the time awake after sleep onset (WASO) will be determined at baseline (sham) and compared after CO2 rebreathing intervention. If the apnea/hypopnea index is improved, the sleep quality is expected to improve accordingly, however, the intervention itself has the potential to disrupt sleep even when only minor changes in CO2 are expected.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Misericordia Medical Centre, Sleep Disorder Centre, Winnipeg, Manitoba
  - Sleep Disorder Centre at Misericordia Health Centre, Winnipeg, Manitoba